CLINICAL TRIAL: NCT05245565
Title: Effects of Modified Precision Functional Sphincter-Preserving Surgery (PPS) on Ultralow Rectal Cancer: A Multicenter Prospective Cohort Study
Brief Title: Effects of Modified Precision Functional Sphincter-Preserving Surgery (PPS) on Ultralow Rectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Feng-Min, Investigator assistant, Shanghai 10th People's Hospital
Other Study IDs: SHSY-IEC-4.1/21-311/01
Record Dates: First submitted 2022-01-28; First posted 2022-02-18 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Rectum Cancer; Stoma Colostomy; Faecal Incontinence; Leakage, Anastomotic
MeSH Terms: conditions — Rectal Neoplasms; Encopresis; Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PPS surgery: Patients who undergo modified PPS surgery in order to preserve anal sphincter function under the premise of radical resection of ultralow rectal cancer.
- Conventional: Patients who undergo conventional sphincter-preserving surgeries.

SUMMARY:
RATIONALE: Colorectal cancer is one of the most common cancers. However, approaches to minimize surgical trauma, preserve anal function, avoid abdominal stoma, and improve quality of life for patients with ultralow rectal cancers were limited. Thus, new technologies are urgently needed to improve the anal preservation rate, reduce the incidence of anastomotic leakage and improve postoperative anal function in patients with ultralow rectal cancer.

PURPOSE: This one-arm multicenter prospective cohort study aims to collect the data of patients with ultralow rectal cancer who undergo sphincter-preserving surgeries, including modified PPS and conventional surgeries, then compare the effects of different operations on clinical outcomes and to see the efficacy and safety of modified PPS surgery when compared with conventional procedures in the treatment of ultralow rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histological proof of newly diagnosed primary adenocarcinoma of the rectum
2. The lower edge of tumor < 3 cm from the dentate line
3. Clinical T stage ≤ T3

Exclusion Criteria:

1. The lower edge of tumor < 1 cm from the dentate line
2. Locally advanced stage of tumor
3. Presence of metastatic disease or recurrent rectal tumor
4. Concomitant malignancies
5. Concurrent uncontrolled medical conditions
6. Impaired anal function before surgery
7. Presence of acute bowel obstruction or bowel perforation caused by cancer
8. Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study population is the patients who diagnosed as low-lying rectal adenocarcinoma cases by preoperative pathology and meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Rate of temporary defunctioning stoma | Within 30 days after operation
  The percentage of patients who get temporary defunctioning stoma to limit the consequences of anastomotic leakage.
The percentage of patients who develop anastomotic leakage | Within 30 days after operation
  The percentage of patients who develop anastomotic leakage
Postoperative anal function assessed by Wexner scale | 2 years since the start of treatment
  Ranging from 0 (perfect continence) to 20 (complete incontinence)
Postoperative anal function assessed by Vaizey scale | 2 years since the start of treatment
  Ranging from 0 (perfect continence) to 24 (complete incontinence)

SECONDARY OUTCOMES:
Rate of sphincter-preservation rates | Within 30 days after operation
  The percentage of patients who preserve the anatomical structure of the anus
The number of short-term postoperative complications | Within 30 days after operation
  The number of grade II and higher postoperative complications according to the Clavien-Dindo classification
Postoperative hospital stay | Within 30 days after operation
  The time between the operation date and the discharge date.
Hospitalization costs | Within 30 days after operation
  The total cost of hospitalization
30-Day Readmission Rate | Within 30 days after operation
  Percentage of readmitted patients within 30 days after operation
Disease-free survival | Up to 5 years after the last patient recruited
  Disease-free survival is defined as the time from surgery to recurrence of tumor or death
Overall survival | Up to 5 years after the last patient recruited
  Overall survival is defined as the time from surgery until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Le Zhuang, MD, PhD, Study Chair — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China